CLINICAL TRIAL: NCT06273241
Title: Impact of Food Intake on Berberine Kinetics - BERKI-3
Brief Title: Impact of Food Intake on Berberine Kinetics
Acronym: BERKI-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Stefan Engeli, MD, Professor, University Medicine Greifswald
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IPHA-2024-009
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Pharmacokinetic Study in Healthy Volunteers
Keywords: berberine; food effect; pharmacokinetic
MeSH Terms: interventions — Eating

STUDY DESIGN:
Intervention Model Description: This is an unblinded, randomized, prospective study comparing berberine intake in fasted condition and after a high or low caloric meal in a cross-over design.
Masking Description: This study will be an open label study. Participants will be selected from an existing database of the Institute of Pharmacology Greifswald.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Berberine intake in fasted condition (Placebo Comparator): Intake of 1000 mg berberine in the fasted condition (intake of last meal: before 20:00 on the day before the study visit)
  Interventions: Other: food intake
- Berberine intake after a low caloric meal (Active Comparator): Intake of 1000 mg berberine after a light caloric meal (2 toasts, butter, cheese, marmalade)
  Interventions: Other: food intake
- Berberine intake after a high caloric meal (Active Comparator): Intake of 1000 mg berberine after a high caloric meal (2 toasts with butter, 2 fried eggs, 2 slices of bacon, 3 hash brown and 240ml of whole milk)
  Interventions: Other: food intake

INTERVENTIONS:
Other: food intake — A single dose of 1000 mg berberine in two capsules will be administered with 250 ml of still water in the overnight fasting condition as the control condition. The two intervention arms will test the effect of different meals on berberine kinetics. A total amount of 12 blood samples at defined time points (baseline; 1; 2; 3; 4; 5; 6; 7; 8; 24 h) will be taken. For glucose and insulin measurements, blood samples will be obtained at 4 h, 5 h and 6 h .

SUMMARY:
The influence of genetic variants of the CYP2D6 enzyme and the Organic Cation Transporter 1 (OCT-1) on the kinetics of berberine (BERKI-1) has recently been studied. A significant sex difference was observed. These results lead to the BERKI-2 study, investigating the influence of the female hormonal cycle on berberine kinetics. In this study, women took a single berberine dose once in the first and once in the second half of their menstrual cycle, men served as a control group ingesting a single berberine dose. Contrary to expectations, the previously observed sex difference could not be confirmed.

In both BERKI-1 and 2 studies, the plasma concentration curve exhibited two peaks. The first after about 2-3 h, and the second after approximately 5 h of berberine intake. All participants took a single dose of Berberine under fasting conditions in the morning and 4 h after berberine intake, the participants ate a meal. Shortly after meal intake, the plasma concentration curve peaked again.

BERKI-3 will investigate the impact of food intake on berberine bioavailability and the kinetic properties. Given the suspected influence of berberine on glycemic control, the investigators will also measure insulin and glucose after the meal at noon.

As in BERKI-1 and 2, time dependent blood and urine samples will be collected after a single berberine dose. One by measuring berberine metabolites by Liquid Chromatography and Mass-spec One dose will be taken in the fasted condition and the other two after a light or high caloric meal, respectively.

24 healthy volunteers with an equal ratio of man and women will be enrolled.

DETAILED DESCRIPTION:
All enrolled participants will come under fasting conditions for 10 h to the Clinical Research Unit. Every volunteer will receive a single dose of 1000 mg berberine (two capsules) with 250 ml still water. Intake will be either in the fasting condition, or after a light caloric meal (2 toasts, butter, cheese, marmalade), or a high caloric meal (2 toasts with butter, 2 fried eggs, 2 slices of bacon, 3 hash brown and 240ml of whole milk), respectively. In between these different intakes will be at least one week. The order of fasting - light meal - heavy meal study visits will be randomized.

A total amount of 12 blood samples at defined time points (baseline; 1; 2; 3; 4; 5; 6; 7; 8; 24 h) will be taken. At each time point, blood will be collected in a tube for collecting plasma. In addition, for glucose and insulin measurements, blood samples will be obtained at 4 h, 5 h and 6 h .

Every hour until the meal at noon, participants will drink 100 ml of sparkling water to stimulate the intestinal peristalsis and promote transport of the capsule. Volunteers are asked to stay in bed for four hours after berberine intake but then are allowed to move freely in the Clinical Research Unit. After 2 h participants will be served tea or coffee and after 4 h a meal will be served.

Urine will be collected at the first 8 h after administration. The participants will stay in the Clinical Research Unit of the Institute of Pharmacology for the first 8 hours after administration.

ELIGIBILITY:
Inclusion Criteria:

* wildtype genotypes for CYP2D6 and organic cation transporter 1 (OCT-1)
* understands the study purpose and design
* contractually capable and provides signed informed consent form
* healthy condition or mild and/or well treated forms of allergies, asthma, hypertension and orthopedic diseases

Exclusion Criteria:

* BMI ≤18,5kg/m2 and ≥29,9 kg/m2
* only in women: known pregnancy or lactation period
* only in women: positive pregnancy test at screening or any other study visit
* anemia: Hb < 13 g/dl (8,07 mmol/l) in men or < 12 g/dl (7,45 mmol/l) in women
* elevated liver function tests (ALAT, ASAT, yGT, Bilirubin > 2xULN)
* reduced renal function (eGFRMDRD < 60ml/min/1,7m2)
* currently mentally unstable
* use of recreational drugs more than twice a week
* poor venous conditions that make it impossible to place a peripheral venous catheter and regularly draw blood through it

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Berberine plasma concentration fasted vs fed | 24 hours
  Difference of berberine plasma concentrations between the fasted and fed condition, expressed as area under the curve (AUC0-24h).

SECONDARY OUTCOMES:
Berberine plasma concentrations light vs heavy meal | 24 hours
  Difference of berberine plasma concentrations after a light and heavy meal, expressed as area under the curve (AUC0-24h).

OTHER OUTCOMES:
Blood glucose concentrations | 2 hours
  AUC of blood glucose over two hours after single doses of berberine, both in the fasted and fed condition.
Blood insulin concentrations | 2 hours
  AUC of blood insulin over two hours after single doses of berberine, both in the fasted and fed condition.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Engeli, Prof., Principal Investigator — Universitätsmedizin Greifswald, Institut für Pharmakologie
Locations (1):
- University Medicine Greifswald, Institute of Pharmacology, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No